CLINICAL TRIAL: NCT01926886
Title: A Single Arm Multi-center Study Investigating the at Home Administration of Trastuzumab Subcutaneous Vial for the Treatment of Patients With HER2-positive Early Breast Cancer
Brief Title: A Study of Subcutaneous At Home Administration of Trastuzumab (Herceptin) in Participants With Human Epidermal Growth Factor Receptor 2-positive (HER2+) Early Breast Cancer (eBC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28794; 2013-000123-13 (EudraCT Number)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (2):
- Trastuzumab (Experimental): Participants with HER2+ eBC who completed the first 6 cycles of trastuzumab IV infusion as part of the (neo) adjuvant treatment will be included to continue to receive 12 cycles of trastuzumab to complete a total of 18 cycles of trastuzumab. Participants will receive trastuzumab IV infusion at initial loading dose of 8 mg/kg BW for q3w regimen as a part of neo adjuvant treatment before entering in the study and then recommended maintenance dose of 6 mg/kg BW q3w for the first 3 cycles (cycles 7-9) in hospital followed by SC administration of trastuzumab at a fixed dose of 600 mg q3w for next 3 cycles (Cycles 10-12) at hospital and SC administration of trastuzumab at a fixed dose of 600 mg q3w at home for the next 6 cycles (Cycles 13-18) (Each cycle=21 days).
  Interventions: Drug: Trastuzumab
- Health Care Professionals (No Intervention): Health Care Professionals (HCPs) included for polling purposes. HCPs were not enrolled in the study.

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab 8 mg/kg (loading dose) and 6 mg/kg (maintenance dose) IV infusion q3w; Trastuzumab 600 mg q3w SC injection will be administered as per the schedule specified in the arm.
  Other Names: Herceptin
  Arms: Trastuzumab

SUMMARY:
This single arm, multicenter study will evaluate the safety of assisted subcutaneous administration of trastuzumab in participants with HER2+ eBC. Participants who have completed the first 6 cycles of intravenous (IV) trastuzumab as part of the (neo)adjuvant treatment will be eligible to receive a further 12 cycles of trastuzumab in this study. Participants will receive IV trastuzumab at initial loading dose of 8 milligrams per kilogram (mg/kg) body weight (BW) for three-weekly (q3w) regimen and then recommended maintenance dose of 6 mg/kg BW q3w for the first 3 cycles (cycles 7-9) in hospital followed by subcutaneous (SC) administration of trastuzumab at a fixed dose of 600 mg q3w for next 3 cycles (Cycles 10-12) at hospital and SC administration of trastuzumab at a fixed dose of 600 mg q3w at home for the next 6 cycles (Cycles 13-18).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast
* HER2-positive disease immunohistochemistry (IHC)3+ or in situ hybridization (ISH) positive, in line with local reimbursement criteria and determined in a local laboratory that is experienced/certified in HER2-expression testing using an accurate and validated assay
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Hormonal therapy will be allowed as per institutional guidelines
* Left ventricular ejection fraction (LVEF) of greater than or equal to (>/=) 50% measured by echocardiography (ECHO) or multiple gated acquisition (MUGA) scan prior to first dose of trastuzumab SC, or, for those who were receiving trastuzumab when beginning the study, documented results within an acceptable limit from a cardiac assessment within 3 months prior to enrollment
* Participants have completed the first 6 cycles of trastuzumab IV as part of the (neo)adjuvant treatment
* No evidence of residual, locally recurrent or metastatic disease after completion of surgery and chemotherapy, (neo-adjuvant or adjuvant)
* Use of concurrent curative radiotherapy will be permitted

Exclusion Criteria:

* History of other malignancy which could affect compliance with the protocol or interpretation of results. Participants with curatively treated carcinoma in situ of the cervix or basal cell carcinoma, and patients with other curatively treated malignancies who have been disease-free for at least 5 years, are eligible
* Participants with severe dyspnea at rest or requiring supplementary oxygen therapy
* Participants with other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness
* Serious cardiac illness or medical conditions that would preclude the use of trastuzumab, specifically: history of documented congestive heart failure (CHF), high-risk uncontrolled arrhythmias, angina pectoris requiring medication, clinically significant valvular disease, evidence of transmural infarction on electrocardiogram (ECG), diagnosed poorly controlled hypertension
* Known infection with human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Pregnant or lactating women
* Women of childbearing potential and male participants with partners of childbearing potential who are unable or unwilling to use adequate contraceptive measures during study treatment
* Concurrent enrollment in another clinical trial using an investigational anti-cancer treatment, including hormonal therapy, bisphosphonate therapy and immunotherapy, within 28 days prior to the first dose of study treatment
* Known hypersensitivity to trastuzumab, murine proteins, to any of the excipients of Herceptin including hyaluronidase, or the adhesive of the SC device, or a history of severe allergic or immunological reactions, e.g. difficult to control asthma
* Inadequate bone marrow, hepatic or renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2015-09-04 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- Belgium (13):
  - Onze Lieve Vrouwziekenhuis Aalst, Aalst
  - Imeldaziekenhuis, Bonheiden
  - AZ Sint Jan, Bruges
  - CHU St Pierre (St Pierre), Brussels
  - AZ Maria Middelares, Ghent
  - AZ Sint Lucas (Sint Lucas), Ghent
  - UZ Gent, Ghent
  - CH Jolimont - Lobbes (Jolimont), Haine-Saint-Paul
  - Clinique Saint-Joseph, Liège
  - CHU Ambroise Paré, Mons
  - CHR de Namur, Namur
  - AZ Damiaan, Ostend
  - AZ Turnhout Sint Elisabeth, Turnhout
- Israel (10):
  - Soroka Medical Center; Oncology Dept, Beersheba
  - Rambam Medical Center; Oncology, Haifa
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Meir Medical Center; Oncology, Kfar Saba
  - Western Galilee Hospital; Oncology-Nahariya, Nahariya
  - Rabin MC; Davidof Center - Oncology Institute, Petah Tikva
  - Chaim Sheba medical center, Oncology division, Ramat Gan
  - Kaplan Medical Center; Oncology Inst., Rehovot
  - Sourasky / Ichilov Hospital; Dept. of Oncology, Tel Aviv
  - Assaf Harofeh; Oncology, Ẕerifin

REFERENCES:
- [Derived] Denys H, Martinez-Mena CL, Martens MT, D'Hondt RG, Graas ML, Evron E, Fried G, Ben-Baruch NE, Vulsteke C, Van Steenberghe MM. Safety and tolerability of subcutaneous trastuzumab at home administration, results of the phase IIIb open-label BELIS study in HER2-positive early breast cancer. Breast Cancer Res Treat. 2020 May;181(1):97-105. doi: 10.1007/s10549-020-05604-7. Epub 2020 Apr 2. PMID 32240454

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with human epidermal growth factor receptor 2-positive (HER2+) early breast cancer (eBC) who completed the first 6 cycles of trastuzumab intravenous (IV) as part of the (neo)adjuvant treatment received 12 cycles of trastuzumab to complete a total of 18 cycles of trastuzumab were enrolled.
Groups:
- Trastuzumab: Participants received trastuzumab IV infusion at initial loading dose of 8 milligrams per kilogram (mg/kg) body weight (BW) for three-weekly (q3w) regimen as a part of neo adjuvant treatment before entering in the study and then recommended maintenance dose of 6 mg/kg BW q3w for the first 3 cycles (Cycles 7-9) in hospital followed by subcutaneous (SC) administration of trastuzumab at a fixed dose of 600 mg q3w for next 3 cycles (Cycles 10-12) at hospital and SC administration of trastuzumab at a fixed dose of 600 mg q3w at home for the next 6 cycles (Cycles 13-18) (Each cycle=21 days).
- Health Care Professionals: HCPs included for polling purposes. HCPs were not enrolled in the study.
Period: Overall Study
Arm/Group | Trastuzumab | Health Care Professionals
Started | 102 | 21 (HCPs were not enrolled in the study. No baseline data were collected for these participants.)
Received at Least 1 Dose of Study Drug | 101 | 0 (Partcipants were HCPs included for polling purposes. HCPs were not enrolled in the study.)
Completed | 70 | 21 (Partcipants were HCPs included for polling purposes. HCPs were not enrolled in the study.)
Not Completed | 32 | 0
Not completed — Administrative/other | 1 | 0
Not completed — Adverse event/intercurrent illness | 4 | 0
Not completed — Disease progression/recurrence | 4 | 0
Not completed — Withdrawal by Subject | 15 | 0
Not completed — Failure to return | 3 | 0
Not completed — Recurrence of disease | 1 | 0
Not completed — Progression of disease | 2 | 0
Not completed — Death | 1 | 0
Not completed — Did not cooperate | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all enrolled participants.
  HCPs included for polling purposes. Baseline information not collected on HCPs. HCPs were not enrolled in the study.
Groups:
- Trastuzumab: Participants received trastuzumab IV infusion at initial loading dose of 8 mg/kg BW for q3w regimen as a part of neo adjuvant treatment before entering in the study and then recommended maintenance dose of 6 mg/kg BW q3w for the first 3 cycles (Cycles 7-9) in hospital followed by SC administration of trastuzumab at a fixed dose of 600 mg q3w for next 3 cycles (Cycles 10-12) at hospital and SC administration of trastuzumab at a fixed dose of 600 mg q3w at home for the next 6 cycles (Cycles 13-18) (Each cycle=21 days).
Arm/Group | Trastuzumab
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.38 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 98
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs included both serious and non- serious AEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An emergent AE was defined as occurring within 35 days after last treatment administration.
Time Frame: Up to 45 months
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 101
percentage of participants
  Emergent AEs | 90.1
  Emergent SAEs | 7.9

2. Secondary Outcome: Number of Participants With Modalities Assessed Using Patient Satisfaction Questionnaire 1 (PSQ1): In-Hospital
Description: PSQ1 is a quality of care questionnaire containing 14 questions each of Sections A and B, with a total of 28 questions categorized on the opinion of participants about the clinicians, opinion of participants about the other staff and other questions. Responses to questions with section A (except question 11) were categorized to "not at all", "to a small extent", "to a moderate extent", "to a large extent", "to a very large extent", "Not applicable" and "missing". Responses to questions with section B were categorized to "Not important", "a little important", "important", "very important", "of utmost importance", "not applicable" and "missing". Responses to question 11 with section A were categorized to "Yes, but not long", "yes, quite long", "yes, much long" and "missing". Participant experience with the treatment provided during the in-hospital part of the study was evaluated with PSQ1 questionnaire completed by the participant prior to the first dose of trastuzumab SC at home.
Time Frame: Prior (0 hour) to first trastuzumab SC administration at Cycle 13 (cycle length =21 days)
Population: ITT population. Here, "number of participants analysed" included participants who were evaluable for the outcome measure.
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 86
participants
  1a:Clinician Communication-Not at all | 0
  1a:Clinician Communication-To a small extent | 4
  1a:Clinician Communication-To a moderate extent | 8
  1a:Clinician Communication-To a large extent | 22
  1a:Clinician Communication-To a very large extent | 49
  1a:Clinician Communication-Not applicable | 0
  1a:Clinician Communication-Missing | 3
  1b:Importance-Not important | 1
  1b:Importance-A little important | 3
  1b:Importance-Important | 19
  1b:Importance-Very important | 40
  1b:Importance-Of utmost importance | 21
  1b:Importance-Not applicable | 0
  1b:Importance-Missing | 2
  2a:Confidence in clinicians-Not at all | 0
  2a:Confidence in clinicians-To a small extent | 0
  2a:Confidence in clinicians-To a moderate extent | 5
  2a:Confidence in clinicians-To a large extent | 23
  2a:Confidence in clinicians-To a very large extent | 56
  2a:Confidence in clinicians-Not Applicable | 0
  2a:Confidence in clinicians-Missing | 2
  2b:Importance-Not important | 0
  2b:Importance-A little important | 1
  2b:Importance-Important | 13
  2b:Importance-Very important | 44
  2b:Importance-Of utmost importance | 25
  2b:Importance-Not applicable | 0
  2b:Importance-Missing | 3
  3a:Clinicians cared about you-Not at all | 2
  3a:Clinicians cared about you-To a small extent | 1
  3a:Clinicians cared about you-To a moderate extent | 6
  3a:Clinicians cared about you-To a large extent | 24
  3a:Clinicians cared about you-To very large extent | 51
  3a:Clinicians cared about you-Not applicable | 0
  3a:Clinicians cared about you-Missing | 2
  3b:Importance-Not important | 0
  3b:Importance-A little important | 2
  3b:Importance-Important | 16
  3b:Importance-Very important | 47
  3b:Importance-Of utmost importance | 18
  3b:Importance-Not applicable | 0
  3b:Importance-Missing | 3
  4a:Clinicians interested-Not at all | 0
  4a:Clinicians interested-To a small extent) | 2
  4a:Clinicians interested-To a moderate extent | 12
  4a:Clinicians interested-To a large extent | 29
  4a:Clinicians interested-To a very large extent | 40
  4a:Clinicians interested-Not applicable | 1
  4a:Clinicians interested-Missing | 2
  4b:Importance-Not important | 0
  4b:Importance-A little important | 2
  4b:Importance-Important | 15
  4b:Importance-Very important | 51
  4b:Importance-Of utmost importance | 15
  4b:Importance-Not applicable | 0
  4b:Importance-Missing | 3
  5a:Time with clinicians-Not at all | 1
  5a:Time with clinicians-To small extent | 4
  5a:Time with clinicians-To a moderate extent | 12
  5a:Time with clinicians-To a large extent | 26
  5a:Time with clinician-To a very large extent | 39
  5a:Time with clinicians-Not applicable | 1
  5a:Time with clinicians-Missing | 3
  5b:Importance-Not important | 0
  5b:Importance-A little important | 2
  5b:Importance-Important | 21
  5b:Importance-Very important | 45
  5b:Importance-Of utmost importance | 14
  5b:Importance-Not applicable | 0
  5b:Importance-Missing | 4
  6a:Nurses communication-Not at all | 0
  6a:Nurses communication-To a small extent | 1
  6a:Nurses communication-To a moderate extent | 4
  6a:Nurses communication-To a large extent | 19
  6a:Nurses communication-To a very large extent | 60
  6a:Nurses communication-Not Applicable | 0
  6a:Nurses communication-Missing | 2
  6b:Importance-Not important | 1
  6b:Importance-A little important | 4
  6b:Importance-Important | 18
  6b:Importance-Very important | 44
  6b:Importance-Of utmost importance | 16
  6b:Importance-Not applicable | 0
  6b:Importance-Missing | 3
  7a:Confidence in nurses-Not at all | 0
  7a:Confidence in nurses-To a small extent | 0
  7a:Confidence in nurses-To a moderate extent | 4
  7a:Confidence in nurses-To a large extent | 19
  7a:Confidence in nurses-To a very large extent | 61
  7a:Confidence in nurses-Not Applicable | 0
  7a:Confidence in nurses-Missing | 2
  7b:Importance-Not important | 0
  7b:Importance-A little important | 1
  7b:Importance-Important | 17
  7b:Importance-Very important | 46
  7b:Importance-Of utmost importance | 19
  7b:Importance-Not applicable | 0
  7b:Importance-Missing | 3
  8a:Nurses cared about you-Not at all | 1
  8a:Nurses cared about you-To a small extent | 2
  8a:Nurses cared about you-To a moderate extent | 4
  8a:Nurses cared about you-To a large extent | 25
  8a:Nurses cared about you-To a very large extent | 52
  8a:Nurses cared about you-Not Applicable | 0
  8a:Nurses cared about you-Missing | 2
  8b:Importance-Not important | 0
  8b:Importance-A little important | 3
  8b:Importance-Important | 22
  8b:Importance-Very important | 41
  8b:Importance-Of utmost importance | 17
  8b:Importance-Not applicable | 0
  8b:Importance-Missing | 3
  9a:Nurses interested-Not at all | 0
  9a:Nurses interested-To a small extent | 3
  9a:Nurses interested-To a moderate extent | 3
  9a:Nurses interested-To a large extent | 22
  9a:Nurses interested-To a very large extent | 56
  9a:Nurses interested-Not Applicable | 0
  9a:Nurses interested-Missing | 2
  9b:Importance-Not important | 0
  9b:Importance-A little important | 5
  9b:Importance-Important | 22
  9b:Importance-Very important | 41
  9b:Importance-Of utmost importance | 14
  9b:Importance-Not applicable | 0
  9b:Importance-Missing | 4
  10a:Time with nurses-Not at all | 0
  10a:Time with nurses-To a small extent | 4
  10a:Time with nurses-To a moderate extent | 10
  10a:Time with nurses-To a large extent | 20
  10a:Time with nurses-To a very large extent | 49
  10a:Time with nurses-Not Applicable | 1
  10a:Time with nurses-Missing | 2
  10b:Importance-Not important | 0
  10b:Importance-A little important | 5
  10b:Importance-Important | 21
  10b:Importance-Very important | 40
  10b:Importance-Of utmost importance | 15
  10b:Importance-Not applicable | 0
  10b:Importance-Missing | 5
  11a:Waited for hospital admission-No | 24
  11aWaited for hospital admission-Yes, but not long | 34
  11a:Waited for hospital admission-Yes, quite long | 20
  11a:Waited for hospital admission-Yes, much long | 4
  11a:Waited for hospital admission-Missing | 4
  11b:Importance-Not important | 5
  11b:Importance-A little important | 12
  11b:Importance-Important | 28
  11b:Importance-Very important | 24
  11b:Importance-Of utmost importance | 12
  11b:Importance-Not applicable | 0
  11b:Importance-Missing | 5
  12a:Clinic equipment good order-Not at all | 0
  12a:Clinic equipment good order-To a small extent | 1
  12a:Clinic equipment good order-To moderate extent | 3
  12a:Clinic equipment good order-To a large extent | 34
  12aClinic equipment good order-To very large exten | 46
  12a:Clinic equipment good order-Not applicable | 0
  12a:Clinic equipment in good order-Missing | 2
  12b:Importance-Not important | 0
  12b:Importance-A little important | 0
  12b:Importance-Important | 22
  12b:Importance-Very important | 41
  12b:Importance-Of utmost importance | 20
  12b:Importance-Not applicable | 0
  12b:Importance-Missing | 3
  13a:Clinic otherwise good order-Not at all | 0
  13a:Clinic otherwise good order-To a small extent | 1
  13a:Clinic otherwise good order-To moderate extent | 5
  13a:Clinic otherwise good order-To a large extent | 32
  13aClinic otherwise good order- Very large extent | 45
  13a:Clinic otherwise good order-Not Applicable | 0
  13a:Clinic otherwise good order-Missing | 3
  13b:Importance-Not important | 0
  13b:Importance-A little important | 2
  13b:Importance-Important | 23
  13b:Importance-Very important | 39
  13b:Importance-Of utmost importance | 18
  13b:Importance-Not applicable | 0
  13b:Importance-Missing | 4
  14a:Satisfactory treatment-Not at all | 0
  14a:Satisfactory treatment-To a small extent | 0
  14a:Satisfactory treatment-To a moderate extent | 1
  14a:Satisfactory treatment-To a large extent | 18
  14a:Satisfactory treatment-To a very large extent | 65
  14a:Satisfactory treatment-Not Applicable | 0
  14a:Satisfactory treatment-Missing | 2
  14b:Importance-Not important | 0
  14b:Importance-A little important | 3
  14b:Importance-Important | 12
  14b:Importance-Very important | 43
  14b:Importance-Of utmost importance | 25
  14b:Importance-Not applicable | 0
  14b:Importance-Missing | 3

3. Secondary Outcome: Number of Participants With Modalities Assessed Using Patient Satisfaction Questionnaire 2 (PSQ2): At Home
Description: PSQ2 is a quality of care questionnaire containing 13 questions each of Sections A and B, with a total of 26 questions categorized on the opinion of participants about the clinicians, opinion of participant about the other staff and other questions. Responses to questions with section A were categorized to "Not at all", "To a small extent", "to a moderate extent", "to a large extent", "to a very large extent", "Not applicable" and "missing". Responses to questions with section B were categorized to "Not important", "a little important", "important", "very important", "of utmost importance", "not applicable" and "missing". Participant experience with the treatment provided during the at-home part of the study was evaluated with the PSQ2 questionnaire completed by the participant prior to the fifth dose of trastuzumab SC at home.
Time Frame: Prior (0 hour) to fifth trastuzumab SC administration at Cycle 17 (cycle length=21 days)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 83
participants
  1a:Clinicians communication-Not at all | 0
  1a:Clinicians communication-To a small extent | 3
  1a:Clinicians communication-To a moderate extent | 8
  1a:Clinicians communication-To a large extent | 28
  1a:Clinicians communication-To a very large extent | 34
  1a:Clinicians communication-Not Applicable | 7
  1a:Clinicians communication-Missing | 3
  1b:Importance-Not important | 2
  1b:Importance-A little important | 0
  1b:Importance-Important | 20
  1b:Importance-Very important | 37
  1b:Importance-Of utmost importance | 16
  1b:Importance-Not applicable | 0
  1b:Importance-Missing | 8
  2a:Confidence in the clinicians-Not at all | 0
  2a:Confidence in the clinicians-To a small extent | 1
  2a:Confidence in the clinicians-To moderate extent | 2
  2a:Confidence in the clinicians-To a large extent | 20
  2a:Confidence in clinician-To very large extent | 51
  2a:Confidence in the clinicians-Not applicable | 5
  2a:Confidence in the clinicians-Missing | 4
  2b:Importance-Not important | 0
  2b:Importance-A little important | 0
  2b:Importance-Important | 14
  2b:Importance-Very important | 38
  2b:Importance-Of utmost importance | 23
  2b:Importance-Not applicable | 0
  2b:Importance-Missing | 8
  3a:Clinicians cared about you-Not at all | 2
  3a:Clinicians cared about you-To a small extent | 1
  3a:Clinicians cared about you-To a moderate extent | 6
  3a:Clinicians cared about you-To a large extent | 22
  3a:Clinician cared about you-To very large extent | 42
  3a:Clinicians cared about you-Not Applicable | 6
  3a:Clinicians cared about you-Missing | 4
  3b:Importance-Not important | 0
  3b:Importance-A little important | 1
  3b:Importance-Important | 20
  3b:Importance-Very important | 34
  3b:Importance-Of utmost importance | 20
  3b:Importance-Not applicable | 0
  3b:Importance-Missing | 8
  4a:Clinicians interested-Not at all | 0
  4a:Clinicians interested-To a small extent | 1
  4a:Clinicians interested-To a moderate extent | 9
  4a:Clinicians interested-To a large extent | 27
  4a:Clinicians interested-To a very large extent | 36
  4a:Clinicians interested-Not applicable | 6
  4a:Clinicians interested-Missing | 4
  4b:Importance-Not important | 0
  4b:Importance-A little important | 1
  4b:Importance-Important | 19
  4b:Importance-Very important | 34
  4b:Importance-Of utmost importance | 21
  4b:Importance-Not applicable | 0
  4b:Importance-Missing | 8
  5a:Clinicians interaction-Not at all | 1
  5a:Clinicians interaction-To a small extent | 0
  5a:Clinicians interaction-To moderate extent | 11
  5a:Clinicians interaction-To a large extent | 31
  5a:Clinicians interaction-To very large extent | 30
  5a:Clinicians interaction-Not Applicable | 6
  5a:Clinicians interaction-Missing | 4
  5b:Importance-Not important | 0
  5b:Importance-A little important | 0
  5b:Importance-Important | 22
  5b:Importance-Very important | 35
  5b:Importance-Of utmost importance | 18
  5b:Importance-Not applicable | 0
  5b:Importance-Missing | 8
  6a:Nurses communication-Not at all | 0
  6a:Nurses communication-To a small extent | 1
  6a:Nurses communication-To a moderate extent | 1
  6a:Nurses communication-To a large extent | 17
  6a:Nurses communication-To a very large extent | 62
  6a:Nurses communication-Not applicable | 1
  6a:Nurses communication-Missing | 1
  6b:Importance-Not important | 0
  6b:Importance-A little important | 0
  6b:Importance-Important | 22
  6b:Importance-Very important | 39
  6b:Importance-Of utmost importance | 21
  6b:Importance-Not applicable | 0
  6b:Importance-Missing | 1
  7a:Confidence in the nurses-Not at all | 0
  7a:Confidence in the nurses-To a small extent | 0
  7a:Confidence in the nurses-To a moderate extent | 1
  7a:Confidence in the nurses-To a large extent | 23
  7a:Confidence in the nurses-To a very large extent | 58
  7a:Confidence in the nurses-Not applicable | 0
  7a:Confidence in the nurses-Missing | 1
  7b:Importance-Not important | 0
  7b:Importance-A little important | 1
  7b:Importance-Important | 17
  7b:Importance-Very important | 41
  7b:Importance-Of utmost importance | 23
  7b:Importance-Not applicable | 0
  7b:Importance-Missing | 1
  8a:Nurses cared about you-Not at all | 0
  8a:Nurses cared about you-To a small extent | 0
  8a:Nurses cared about you-To a moderate extent | 2
  8a:Nurses cared about you-To a large extent | 23
  8a:Nurses cared about you-To a very large extent | 57
  8a:Nurses cared about you-Not applicable | 0
  8a:Nurses cared about you-Missing | 1
  8b:Importance-Not important | 0
  8b:Importance-A little important | 1
  8b:Importance-Important | 22
  8b:Importance-Very important | 38
  8b:Importance-Of utmost importance | 20
  8b:Importance-Not applicable | 0
  8b:Importance-Missing | 2
  9a:Nurses interested-Not at all | 0
  9a:Nurses interested-To a small extent | 0
  9a:Nurses interested-To a moderate extent | 4
  9a:Nurses interested-To a large extent | 29
  9a:Nurses interested-To a very large extent | 49
  9a:Nurses interested-Not applicable | 0
  9a:Nurses interested-Missing | 1
  9b:Importance-Not important | 0
  9b:Importance-A little important | 2
  9b:Importance-Important | 27
  9b:Importance-Very important | 34
  9b:Importance-Of utmost importance | 18
  9b:Importance-Not applicable | 0
  9b:Importance-Missing | 2
  10a:Nurses interaction-Not at all | 0
  10a:Nurses interaction-To a small extent | 1
  10a:Nurses interaction-To a moderate extent | 6
  10a:Nurses interaction-To a large extent | 26
  10a:Nurses interaction-To a very large extent | 49
  10a:Nurses interaction-Not applicable | 0
  10a:Nurses interaction-Missing | 1
  10a:Importance-Not important | 0
  10a:Importance-A little important | 3
  10b:Importance-Important | 27
  10b:Importance-Very important | 34
  10b:Importance-Of utmost importance | 17
  10b:Importance-Not applicable | 0
  10b:Importance-Missing | 2
  11a:Nurses equipment good order-Not at all | 0
  11a:Nurses equipment good order-To a small extent | 0
  11a:Nurses equipment good order-To moderate extent | 2
  11a:Nurses equipment good order-To a large extent | 27
  11a:Nurse equipment good order-To verylarge extent | 51
  11a:Nurses equipment good order-Not applicable | 1
  11a:Nurses equipment good order-Missing | 2
  11b:Importance-Not important | 1
  11b:Importance-A little important | 2
  11b:Importance-Important | 21
  11b:Importance-Very important | 41
  11b:Importance-Of utmost importance | 17
  11b:Importance-Not applicable | 0
  11b:Importance-Missing | 1
  12a:Satisfaction-Not at all | 0
  12a:Satisfaction-To a small extent | 0
  12a:Satisfaction-To a moderate extent | 0
  12a:Satisfaction-To a large extent | 14
  12a:Satisfaction-To a very large extent | 67
  12a:Satisfaction-Not applicable | 0
  12a:Satisfaction-Missing | 2
  12a:Importance-Not important | 0
  12a:Importance-A little important | 0
  12b:Importance-Important | 18
  12b:Importance-Very important | 42
  12b:Importance-Of utmost importance | 22
  12b:Importance-Not applicable | 0
  12b:Importance-Missing | 1
  13a:Care benefit at home-Not at all | 0
  13a:Care benefit at home-To a small extent | 0
  13a:Care benefit at home-To moderate extent | 0
  13a:Care benefit at home-To a large extent | 18
  13a:Care benefit at home-To very large extent | 63
  13a:Care benefit at home-Not applicable | 0
  13a:Care benefit at home-Missing | 2
  13b:Importance-Not important | 0
  13b:Importance-A little important | 1
  13b:Importance-Important | 19
  13b:Importance-Very important | 41
  13b:Importance-Of utmost importance | 21
  13b:Importance-Not applicable | 0
  13b:Importance-Missing | 1

4. Secondary Outcome: Participant-reported Severity of Symptoms as Assessed by Monroe Dunaway Anderson Symptom Inventory (MDASI) Questionnaire
Description: MDASI questionnaire is used to rate the severity of 13 core items (pain, fatigue, nausea, vomiting, disturbed sleep, distress, shortness of breath, memory difficulties, lack of appetite, drowsiness, dry mouth, sadness, numbness or tingling). Participants were asked to rate the severity of each symptom "at its worst" using 0-10 numerical rating scales with 0 = "not present" and 10 = "as bad as you can imagine." Total score was summed and ranged from 0 to 130, with lower scores indicating better outcome.
Time Frame: Prior (0 hours) to Cycles 7, 10, 13, 16 (Each cycle=21 days)
Population: ITT population. Here, "number of participants analysed" included participants who were evaluable for the outcome measure and "n" included participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 101
units on a scale
  Pain- IV (Hospital) - Cycle 7 | 1.79 (2.51)
  Fatigue- IV (Hospital) - Cycle 7 | 3.76 (2.69)
  Nausea- IV (Hospital) - Cycle 7: number analyzed (Participants) | 99
  Nausea- IV (Hospital) - Cycle 7 | 0.82 (1.96)
  Disturbed Sleep- IV (Hospital) - Cycle 7 | 3.01 (2.89)
  Distressed- IV (Hospital) - Cycle 7 | 1.99 (2.27)
  Breath shortness- IV (Hospital) - Cycle 7 | 1.59 (2.13)
  Remembering things-IV (Hospital) - Cycle 7: number analyzed (Participants) | 100
  Remembering things-IV (Hospital) - Cycle 7 | 1.97 (2.32)
  Lack of appetite-IV (Hospital) - Cycle 7 | 0.85 (1.80)
  Drowsy- IV (Hospital) - Cycle 7 | 2.25 (2.54)
  Dry mouth- IV (Hospital) - Cycle 7 | 1.89 (2.51)
  Feeling sad- IV (Hospital) - Cycle 7: number analyzed (Participants) | 100
  Feeling sad- IV (Hospital) - Cycle 7 | 1.90 (2.26)
  Vomiting- IV (Hospital) - Cycle 7 | 0.34 (1.31)
  Numbness- IV (Hospital) - Cycle 7 | 3.01 (3.20)
  Pain- SC (Hospital) - Cycle 10: number analyzed (Participants) | 88
  Pain- SC (Hospital) - Cycle 10 | 1.81 (2.14)
  Fatigue- SC (Hospital) - Cycle 10: number analyzed (Participants) | 89
  Fatigue- SC (Hospital) - Cycle 10 | 3.35 (2.45)
  Nausea- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Nausea- SC (Hospital) - Cycle 10 | 0.61 (1.41)
  Disturbed Sleep- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Disturbed Sleep- SC (Hospital) - Cycle 10 | 2.70 (2.86)
  Distressed- SC (Hospital) - Cycle 10: number analyzed (Participants) | 89
  Distressed- SC (Hospital) - Cycle 10 | 2.10 (2.57)
  Breath shortness- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Breath shortness- SC (Hospital) - Cycle 10 | 1.29 (1.88)
  Remembering thing- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Remembering thing- SC (Hospital) - Cycle 10 | 2.01 (2.21)
  Lack of appetite- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Lack of appetite- SC (Hospital) - Cycle 10 | 0.81 (1.67)
  Drowsy- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Drowsy- SC (Hospital) - Cycle 10 | 2.32 (2.52)
  Dry mouth- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Dry mouth- SC (Hospital) - Cycle 10 | 1.42 (2.06)
  Feeling sad- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Feeling sad- SC (Hospital) - Cycle 10 | 1.87 (2.38)
  Vomiting- SC (Hospital) - Cycle 10: number analyzed (Participants) | 89
  Vomiting- SC (Hospital) - Cycle 10 | 0.26 (0.81)
  Numbness- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Numbness- SC (Hospital) - Cycle 10 | 2.73 (2.76)
  Pain- SC (Home) - Cycle 13: number analyzed (Participants) | 83
  Pain- SC (Home) - Cycle 13 | 1.54 (2.33)
  Fatigue- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Fatigue- SC (Home) - Cycle 13 | 3.42 (2.27)
  Nausea- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Nausea- SC (Home) - Cycle 13 | 0.45 (1.25)
  Disturbed Sleep- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Disturbed Sleep- SC (Home) - Cycle 13 | 2.63 (2.50)
  Distressed- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Distressed- SC (Home) - Cycle 13 | 1.81 (2.27)
  Breath shortness- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Breath shortness- SC (Home) - Cycle 13 | 1.28 (2.06)
  Remembering things- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Remembering things- SC (Home) - Cycle 13 | 1.95 (2.07)
  Lack of appetite- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Lack of appetite- SC (Home) - Cycle 13 | 0.43 (1.29)
  Drowsy- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Drowsy- SC (Home) - Cycle 13 | 1.87 (2.26)
  Dry mouth- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Dry mouth- SC (Home) - Cycle 13 | 1.57 (2.30)
  Feeling sad- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Feeling sad- SC (Home) - Cycle 13 | 1.80 (2.32)
  Vomiting- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Vomiting- SC (Home) - Cycle 13 | 0.22 (1.16)
  Numbness- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Numbness- SC (Home) - Cycle 13 | 2.51 (2.64)
  Pain- SC (Home) - Cycle 16: number analyzed (Participants) | 83
  Pain- SC (Home) - Cycle 16 | 1.49 (2.06)
  Fatigue- SC (Home) - Cycle 16: number analyzed (Participants) | 84
  Fatigue- SC (Home) - Cycle 16 | 2.79 (2.05)
  Nausea- SC (Home) - Cycle 16: number analyzed (Participants) | 83
  Nausea- SC (Home) - Cycle 16 | 0.57 (1.35)
  Disturbed Sleep- SC (Home) - Cycle 16: number analyzed (Participants) | 83
  Disturbed Sleep- SC (Home) - Cycle 16 | 2.11 (2.28)
  Distressed- SC (Home) - Cycle 16: number analyzed (Participants) | 84
  Distressed- SC (Home) - Cycle 16 | 2.01 (2.33)
  Breath shortness- SC (Home) - Cycle 16: number analyzed (Participants) | 84
  Breath shortness- SC (Home) - Cycle 16 | 1.38 (2.05)
  Remembering things- SC (Home) - Cycle 16: number analyzed (Participants) | 84
  Remembering things- SC (Home) - Cycle 16 | 2.14 (2.12)
  Lack of appetite- SC (Home) - Cycle 16: number analyzed (Participants) | 84
  Lack of appetite- SC (Home) - Cycle 16 | 0.71 (1.63)
  Drowsy- SC (Home) - Cycle 16: number analyzed (Participants) | 84
  Drowsy- SC (Home) - Cycle 16 | 1.74 (2.01)
  Dry mouth- SC (Home) - Cycle 16: number analyzed (Participants) | 84
  Dry mouth- SC (Home) - Cycle 16 | 1.39 (1.93)
  Feeling sad- SC (Home) - Cycle 16: number analyzed (Participants) | 84
  Feeling sad- SC (Home) - Cycle 16 | 1.98 (2.24)
  Vomiting- SC (Home) - Cycle 16: number analyzed (Participants) | 83
  Vomiting- SC (Home) - Cycle 16 | 0.14 (0.61)
  Numbness- SC (Home) - Cycle 16: number analyzed (Participants) | 84
  Numbness- SC (Home) - Cycle 16 | 2.00 (2.29)

5. Secondary Outcome: Participant-reported Interference of Symptoms With Life as Assessed by MDASI Questionnaire
Description: MDASI questionnaire is used to rate the interference of symptoms. The measure includes 6 symptom interference items which ask how much all symptoms, interfere with domains (general activity, mood, work, relations with others, walking, and enjoyment of life). Each items were rated on a 0-10 scale (0 = "did not interfere"; 10 = "interfered completely"). Lower scores indicating better outcome. Total score was summed and ranged from 0 to 50, with lower scores indicating better outcome.
Time Frame: Prior (0 hours) to Cycles 7, 10, 13, 16 (Each cycle=21 days)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trastuzumab
Number analyzed (Participants) | 101
units on a scale
  General activity- IV (Hospital) - Cycle 7 | 2.77 (2.73)
  Mood- IV (Hospital) - Cycle 7 | 2.11 (2.13)
  Work- IV (Hospital) - Cycle 7 | 3.22 (2.86)
  Relations- IV (Hospital) - Cycle 7 | 1.54 (2.13)
  Walking- IV (Hospital) - Cycle 7: number analyzed (Participants) | 99
  Walking- IV (Hospital) - Cycle 7 | 3.34 (3.06)
  Enjoyment of life- IV (Hospital) - Cycle 7 | 2.51 (2.55)
  General activity- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  General activity- SC (Hospital) - Cycle 10 | 2.24 (2.35)
  Mood- SC (Hospital) - Cycle 10: number analyzed (Participants) | 89
  Mood- SC (Hospital) - Cycle 10 | 1.92 (2.28)
  Work- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Work- SC (Hospital) - Cycle 10 | 2.63 (2.71)
  Relations- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Relations- SC (Hospital) - Cycle 10 | 1.48 (2.30)
  Walking- SC (Hospital) - Cycle 10: number analyzed (Participants) | 89
  Walking- SC (Hospital) - Cycle 10 | 2.38 (2.69)
  Enjoyment of life- SC (Hospital) - Cycle 10: number analyzed (Participants) | 90
  Enjoyment of life- SC (Hospital) - Cycle 10 | 2.21 (2.67)
  General activity- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  General activity- SC (Home) - Cycle 13 | 2.27 (2.48)
  Mood- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Mood- SC (Home) - Cycle 13 | 1.81 (2.28)
  Work- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Work- SC (Home) - Cycle 13 | 2.35 (2.26)
  Relations- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Relations- SC (Home) - Cycle 13 | 1.13 (1.93)
  Walking- SC (Home) - Cycle 13: number analyzed (Participants) | 85
  Walking- SC (Home) - Cycle 13 | 2.13 (2.79)
  Enjoyment of life- SC (Home) - Cycle 13: number analyzed (Participants) | 86
  Enjoyment of life- SC (Home) - Cycle 13 | 2.06 (2.66)
  General activity- SC (Home) - Cycle 16: number analyzed (Participants) | 82
  General activity- SC (Home) - Cycle 16 | 1.84 (2.12)
  Mood- SC (Home) - Cycle 16: number analyzed (Participants) | 82
  Mood- SC (Home) - Cycle 16 | 1.76 (2.13)
  Work- SC (Home) - Cycle 16: number analyzed (Participants) | 83
  Work- SC (Home) - Cycle 16 | 2.00 (2.21)
  Relations- SC (Home) - Cycle 16: number analyzed (Participants) | 82
  Relations- SC (Home) - Cycle 16 | 1.02 (1.85)
  Walking- SC (Home) - Cycle 16: number analyzed (Participants) | 83
  Walking- SC (Home) - Cycle 16 | 1.67 (2.41)
  Enjoyment of life- SC (Home) - Cycle 16: number analyzed (Participants) | 83
  Enjoyment of life- SC (Home) - Cycle 16 | 1.90 (2.37)

6. Secondary Outcome: Number of Participants With Modalities Assessed Using Patient Experience Questionnaires (PEX) - Part 1:In-Hospital
Description: PEX-Part 1 questionnaire contains 25 items to assess participant's experience on use of trastuzumab at hospital.1.Place of treatment? 2.Was it same place as for chemotherapy? 3.How long did it take to travel there? 4.How easy was travel? 5.Company required for travelling? 6.Was travelling cost a problem? 7.Considering all these,was travelling for treatment overall a problem? 8.How helpful were nursing/medical staff? 9.How pleasant was place of study? 10.How was IV treatment given? 11.If Venous Access Device(VAD),what was it? 12.Did hospital staff have difficulty inserting cannula? 13.Time for cannulation? 14.How painful was IV? 15.How much time to access port/line usually take? 16.How painful was it? 17.Time for IV sessions? 18.Anxiety level while IV treatment? 19.How would you describe IV sessions? 20.Did hospital staff have difficulty giving SC? 21.Time for SC? 22.How painful was SC? 23.Time for SC sessions? 24.Anxiety level while SC treatment? 25.How would you describe SC sessions?
Time Frame: Prior (0 hours) to Cycle 12 (cycle length=21 days)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 102
participants
  Place of study treatment: hospital chemo dept | 87
  Place of study treatment: other chemo clinic | 0
  Place of study treatment: Doctor's office | 0
  Place of study treatment: other | 0
  Place of study treatment: missing | 15
  Same place as for your chemotherapy: yes | 87
  Same place as for your chemotherapy: no | 0
  Same place as for your chemotherapy: missing | 15
  Travel time: <1 hour | 70
  Travel time: 1 to 2 hours | 12
  Travel time: >2 hours | 5
  Travel time: missing | 15
  Travelling easy: not at all | 9
  Travelling easy: fairly | 44
  Travelling easy: very | 34
  Travelling easy: missing | 15
  Company required for travelling: always | 32
  Company required for travelling: sometimes | 19
  Company required for travelling: never | 36
  Company required for travelling: missing | 15
  Travelling cost, a problem: not at all | 60
  Travelling cost, a problem: fairly | 23
  Travelling cost, a problem: very | 4
  Travelling cost, a problem: missing | 15
  Travelling overall, a problem: yes | 18
  Travelling overall, a problem: no | 69
  Travelling overall, a problem: missing | 15
  Nursing and medical staff helpful: not at all | 0
  Nursing and medical staff helpful: fairly | 15
  Nursing and medical staff helpful: very | 72
  Nursing and medical staff helpful: missing | 15
  Pleasant place of treatment: not at all | 3
  Pleasant place of treatment: fairly | 39
  Pleasant place of treatment: very | 44
  Pleasant place of treatment: missing | 16
  IV administration method: cannula/needle | 34
  IV administration method:Venous Access Device(VAD) | 47
  IV administration method: both | 6
  IV administration method: missing | 15
  VAD: Hickman | 0
  VAD: peripherally inserted central catheters | 5
  VAD: port-a-cath | 47
  VAD: other | 9
  VAD: missing | 41
  Difficulty inserting the cannula: very often | 5
  Difficulty inserting the cannula: sometimes | 15
  Difficulty inserting the cannula: never | 22
  Difficulty inserting the cannula: missing | 60
  Time for insertion of the cannula: <5 minutes | 30
  Time for insertion of the cannula: 6-10 minutes | 7
  Time for insertion of the cannula: 11-15 minutes | 1
  Time for insertion of the cannula:16-20 minutes | 0
  Time for insertion of the cannula: >20 minutes | 2
  Time for insertion of the cannula: missing | 62
  Cannulation painfull: not at all | 20
  Cannulation painfull: fairly | 18
  Cannulation painfull: very | 4
  Cannulation painfull: missing | 60
  Time for connection to the access port: <5 minutes | 39
  Time for connection to access port: 6-10 minutes | 8
  Time for connection to access port: 11-15 minutes | 1
  Time for connection to access port: 16-20 minutes | 1
  Time for connection to access port: >20 minutes | 0
  Time for connection to access port: missing | 53
  Connection painful: not at all | 36
  Connection painful: fairly | 14
  Connection painful: very | 0
  Connection painful: missing | 52
  Time for IV session: <2 hours | 21
  Time for IV session: 2-3 hours | 25
  Time for IV session: 3-4 hours | 26
  Time for IV session: >4 hours | 13
  Time for IV session: missing | 17
  Anxiety during IV treatment: not at all | 64
  Anxiety during IV treatment: fairly | 20
  Anxiety during IV treatment: very | 2
  Anxiety during IV treatment: missing | 16
  General IV session: very unpleasant | 2
  General IV session: fairly unpleasant | 15
  General IV session: acceptable | 68
  General IV session: missing | 17
  Difficulty in SC injection: very often | 0
  Difficulty in SC injection: sometimes | 4
  Difficulty in SC injection: never | 82
  Difficulty in SC injection: missing | 16
  Time for SC injection: <5 minutes | 56
  Time for SC injection: 6-10 minutes | 26
  Time for SC injection: 11-15 minutes | 1
  Time for SC injection: 16-20 minutes | 0
  Time for SC injection: >20 minutes | 3
  Time for SC injection: missing | 16
  SC injection painful: not at all | 53
  SC injection painful: fairly | 33
  SC injection painful: very | 1
  SC injection painful: missing | 15
  Time for SC session: <2 hours | 46
  Time for SC session: 2-3 hours | 24
  Time for SC session: 3-4 hours | 9
  Time for SC session: >4 hours | 7
  Time for SC session: missing | 16
  Anxiety during SC treatment: not at all | 63
  Anxiety during SC treatment: fairly | 21
  Anxiety during SC treatment: very | 3
  Anxiety during SC treatment: missing | 15
  General SC session: very unpleasant | 0
  General SC session: fairly unpleasant | 7
  General SC session: acceptable | 79
  General SC session: missing | 16

7. Secondary Outcome: Number of Participants With Modalities Assessed Using PEX - Part 2: At Home
Description: PEX - Part 2 questionnaire contains 6 items to assess the participant's experience on the use of trastuzumab SC vials at home.Participants answered the following questions: 1. Did the nursing staff ever have any difficulty giving the trastuzumab injection SC? 2. How many minutes did the injection (it) usually take? 3. How painful was this usually? 4. How long did the SC sessions usually last from arrival until departure of the nurse? 5. How anxious did having the SC treatment make you feel? 6. In general how would you describe these SC treatment sessions at home?
Time Frame: 1 month after end of treatment (up to 10 months)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 102
participants
  Difficulty in SC administration: very often | 0
  Difficulty in SC administration: sometimes | 5
  Difficulty in SC administration: never | 77
  Difficulty in SC administration: missing | 20
  SC administration time: <5 minutes | 65
  SC administration time: 6-10 minutes | 17
  SC administration time: 11-15 minutes | 0
  SC administration time: 16-20 minutes | 0
  SC administration time: >20 minutes | 0
  SC administration time: missing | 20
  SC administration Painful: not at all | 61
  SC administration Painful: fairly | 20
  SC administration Painful: very | 0
  SC administration Painful: missing | 21
  Time for SC session: <2 hours | 82
  Time for SC session: 2-3 hours | 0
  Time for SC session: 3-4 hours | 0
  Time for SC session: >4 hours | 0
  Time for SC session: missing | 20
  Anxiety during SC treatment: not at all | 71
  Anxiety during SC treatment: fairly | 11
  Anxiety during SC treatment: very | 0
  Anxiety during SC treatment: missing | 20
  General SC session: very unpleasant | 3
  General SC session: fairly unpleasant | 0
  General SC session: acceptable | 79
  General SC session: missing | 20

8. Secondary Outcome: Number of Health Care Professionals With Modalities Assessed Using Health Care Professional Questionnaire (HCPEX-1)
Description: HCPEX-1 questionnaire is used to assess health care professional's overall satisfaction and perceived time savings with trastuzumab SC vial in the hospital. The HCPEX-1 questionnaire (19 questions) was completed by the health care professionals administering the trastuzumab IV and SC in the hospital after at least 3 participants had completed the in-hospital part of the study.
Time Frame: Prior (0 hours) to Cycle 12 (cycle length=21 days)
Population: Health care professionals who participated in the study and completed the HCPEX-1 questionnaire.
Measure: Number; unit: Health care professionals
Arm/Group | Health Care Professionals
Number analyzed (Participants) | 21
Health care professionals
  Specialty: Oncologist | 0
  Specialty: Gynecologist | 0
  Specialty: Oncologist/ Specialist Chemo Nurse | 19
  Specialty: Other | 2
  Specialty: Missing | 0
  Personal administration of SC: always | 6
  Personal administration of SC: sometimes | 15
  Personal administration of SC: never | 0
  Personal administration of SC: missing | 0
  Time required for SC preparation: <5 minutes | 7
  Time required for SC preparation: 6-10 minutes | 2
  Time required for SC preparation: 11-15 minutes | 1
  Time required for SC preparation: 16-20 minutes | 1
  Time required for SC preparation: >20 minutes | 1
  Time required for SC preparation: not sure | 9
  Time required for SC preparation: missing | 0
  Time required for SC administration: <3 minutes | 1
  Time required for SC administration: <5 minutes | 16
  Time required for SC administration: 6-15 minutes | 3
  Time required for SC administration: 16-30 minutes | 1
  Time required for SC administration: 31-60 minutes | 0
  Time required for SC administration: 61-90 minutes | 0
  Time required for SC administration: >90 minutes | 0
  Time required for SC administration: not sure | 0
  Time required for SC administration: missing | 0
  Time for SC session: <2 hours | 14
  Time for SC session: 2-3 hours | 7
  Time for SC session: 3-4 hours | 0
  Time for SC session: >4 hours | 0
  Time for SC session: missing | 0
  Reliability of SC hand held syringe: not at all | 0
  Reliability of SC hand held syringe: fairly | 10
  Reliability of SC hand held syringe: very | 11
  Reliability of SC hand held syringe: missing | 0
  Easy to administer SC hand held syringe:not at all | 0
  Easy to administer SC hand held syringe: fairly | 13
  Easy to administer SC hand held syringe: very | 8
  Easy to administer SC hand held syringe: missing | 0
  convenient method for IV treatment- cannula | 7
  convenient method for IV treatment- VAD | 14
  convenient method for IV treatment- not sure | 0
  convenient method for IV treatment- missing | 0
  Personally administer IV: always | 4
  Personally administer IV: sometimes | 15
  Personally administer IV: never | 2
  Personally administer IV: missing | 0
  Personally Cannulate: always | 5
  Personally Cannulate: sometimes | 10
  Personally Cannulate: never | 5
  Personally Cannulate: missing | 1
  Time for IV preparation: <5 minutes | 1
  Time for IV preparation: 6-10 minutes | 2
  Time for IV preparation: 11-15 minutes | 2
  Time for IV preparation: 16-20 minutes | 1
  Time for IV preparation: >20 minutes | 5
  Time for IV preparation: not sure | 10
  Time for IV preparation: missing | 0
  Time for cannulation: <5 minutes | 8
  Time for cannulation: 6-10 minutes | 4
  Time for cannulation: 11-15 minutes | 1
  Time for cannulation: 16-20 minutes | 0
  Time for cannulation: >20 minutes | 2
  Time for cannulation: not sure | 5
  Time for cannulation: missing | 1
  Time for connection: <3 minutes | 1
  Time for connection: <5 minutes | 3
  Time for connection: 6-15 minutes | 0
  Time for connection: 16-30 minutes | 2
  Time for connection: 31-60 minutes | 8
  Time for connection: 61-90 minutes | 5
  Time for connection: >90 minutes | 1
  Time for connection: not sure | 1
  Time for connection: missing | 0
  Time for IV session: <2 hours | 5
  Time for IV session: 2-3 hours | 11
  Time for IV session: 3-4 hours | 4
  Time for IV session: >4 hours | 1
  Time for IV session: missing | 0
  Anxiety during IV treatment: not at all | 14
  Anxiety during IV treatment: fairly | 6
  Anxiety during IV treatment: very | 1
  Anxiety during IV treatment: missing | 0
  Reliablily of IV treatment: not at all | 0
  Reliablily of IV treatment: fairly | 8
  Reliablily of IV treatment: very | 13
  Reliablily of IV treatment: missing | 0
  IV administration easy: not at all | 0
  IV administration easy: fairly | 12
  IV administration easy: very | 9
  IV administration easy: missing | 0
  Quickest administration: IV | 0
  Quickest administration: SC (handheld syringe) | 21
  Quickest administration: no difference | 0
  Quickest administration: missing | 0
  Require less resource: IV | 0
  Require less resource: SC (handheld syringe) | 21
  Require less resource: no difference | 0
  Require less resource: missing | 0

9. Secondary Outcome: Disease-Free Survival (DFS) as Assessed by Routine Clinical, Radiological and Laboratory Criteria
Description: DFS was defined as time from first study drug administration (i.e. Day 1 of Cycle 7) to local, regional or distant recurrence, contralateral breast cancer or death from any cause (whichever occurred first). Diagnosis of breast cancer relapse was made based on routine clinical, radiological and laboratory criteria. Acceptable methods of confirmation of recurrence included radiology, computerized tomography (CT) scan, brain scan, ultrasound, or cytology, as per local practice. In case of uncertainly, disease relapse was to be confirmed by histological or cytological examination of a suspicious lesion, if possible.
Time Frame: From start of treatment up to 45 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab
Number analyzed (Participants) | 102
months | NA [NA to NA] — Median and 95% CI could not be calculated due to low number of events.

ADVERSE EVENTS:
Time Frame: Up to 45 months
Description: An emergent adverse event was defined as occurring within 35 days after last treatment administration. Safety Population
Arm/Group | Trastuzumab | Health Care Professionals
All-Cause Mortality (participants affected / at risk) | 2/101 | 0/0
Serious Adverse Events (participants affected / at risk) | 8/101 | 0/0
Other Adverse Events (participants affected / at risk) | 44/101 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=101) | Health Care Professionals (N=0)
Vertigo (Ear and labyrinth disorders) | 1 | NA
Infected lymphocele (Infections and infestations) | 1 | NA
Ejection fraction decreased (Investigations) | 5 | NA
Lymphoedema (Vascular disorders) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=101) | Health Care Professionals (N=0)
Fatigue (General disorders) | 34 | 0
Injection site erythema (General disorders) | 14 | 0
Injection site swelling (General disorders) | 14 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT01926886/Prot_SAP_000.pdf